CLINICAL TRIAL: NCT04042012
Title: Effect of the Application of Ultrasound-guided Percutaneous Needle Electrolysis on the Chronic Soleus Injury in Dancers
Brief Title: Percutaneous Needle Electrolysis (PNE) in Soleus Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Blanca de la Cruz Torres, Principal investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNE in soleus
Record Dates: First submitted 2019-07-27; First posted 2019-08-01 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Soleus Injury

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eccentric group (Experimental): The dancers of this group wil perform a soleus eccentric exercise
  Interventions: Other: Eccentric exercise
- PNE group (Experimental): The dancers of this group will receive a PNE treatment, consisting of the application of galvanic current, by ultrasound.
  The approach will be performed with a transverse axis with a needle orientation that will depend on the location of the target tissue. The parameters will be 3 mA, 3 seconds, 3 impacts (3: 3: 3). The periodicity will be 1day/7day/21day
  Interventions: Other: PNE
- Combined group (Experimental): The dancers of this group will receive a combined treatment and will be carried out in the same way as the other two groups.
  Interventions: Other: Combined

INTERVENTIONS:
Other: Eccentric exercise — soleus eccentric exercise
  Arms: Eccentric group
Other: PNE — the application of galvanic current
  Arms: PNE group
Other: Combined — soleus eccentric exercise and PNE
  Arms: Combined group

SUMMARY:
This study evaluates if the physiotherapy treatment based on eccentric exercise, ultrasound-guided PNE or a combination of both therapies on chronic soleous injuries may cause changes in pain, functionality, dorsal flexion of the foot, balance and muscle fatigue in dancers.

ELIGIBILITY:
Inclusion Criteria:

* Over 16 years.
* at least 5 years of formal dance training.
* at least 20 hours of training per week.
* Pain in the back of the leg
* diagnosis of chronic soleus injury

Exclusion Criteria:

* Unsurpassed fear of needles
* History of adverse reactions to needles
* Immune system disorder
* Difficulty expressing your feelings properly
* Epilepsy and / or allergies to metals.
* Other lower limbs pathology

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
change of pain level | Change from Baseline VAS at 3 months months
  Visual Analogue Scale (VAS: 0=no pain; 100= pain as bad as can be
Change of Lunge Test | Change from Baseline lunge test at 3 months months
  This test measures the ankle range of motion. Less than 9/10 cm, range of motion will be considered restricted
Change of the Releve test | Change from Baseline releve test at 3 months months
  During the unilateral balance test with open eyes, the participant will be asked to hold as much time as possible in the relay position (raised heel of the floor) on one leg
Change of the Endurance test | Change from Baseline endurance test at 3 months months
  The unilateral raised heel test. The dancer should repeatedly lift the heel from the floor to the maximum range of plantar flexion movement as many times as possible.
Change of the Balance test | Change from Baseline balance test at 3 months months
  The test will be conducted with closed eyes, flat feet and barefoot participants and dancers will perform a retiré position. Participants will maintain the position as long as possible.
Changes of the DFOS questionnaire | Change from Baseline DFOS questionnaire at 3 months months
  This questionnaire measures the pain and function (0= bad; 90=well)
Change of the Minimal Detectable Change (MCD) | Change from after treatment at 3 months months
  The minimal detectable change is defined as a valid change in score that is not due to chance. Minimally clinically important difference (MCID), in comparison, goes beyond valid change to assess meaningful difference in dance function

CONTACTS AND LOCATIONS:
Locations (1):
- University of Seville, Seville, Spain

REFERENCES:
- [Derived] De-la-Cruz-Torres B, Barrera-Garcia-Martin I, Valera-Garrido F, Minaya-Munoz F, Romero-Morales C. Ultrasound-Guided Percutaneous Needle Electrolysis in Dancers with Chronic Soleus Injury: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2020 Aug 27;2020:4156258. doi: 10.1155/2020/4156258. eCollection 2020. PMID 32908559